CLINICAL TRIAL: NCT04809064
Title: Open Versus Arthroscopic Stabilization of Shoulder Instability With Subcritical Bone Loss: The OASIS Trial
Acronym: OASIS
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Adam Popchak, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY21010135; W81XWH-19-PROP-CTA (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Dislocation; Glenohumeral Dislocation; Anterior Shoulder Dislocation
Keywords: Anterior Shoulder Instability; Glenoid Bone Loss; Stabilization Surgery; Return to Duty or Sport; Rehabilitation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Arthroscopic Bankart repair with remplissage of Hill-Sachs lesion/rehabilitation: Arthroscopic Bankart repair surgery with remplissage of Hill-Sachs lesion and post-operative rehabilitation.
  Interventions: Procedure: Arthroscopic Bankart repair procedure; Other: Post-Operative Rehabilitation
- Open Bankart/rehabilitation: Open Bankart surgery and post-operative rehabilitation.
  Interventions: Procedure: Open Bankart; Other: Post-Operative Rehabilitation
- Latarjet/rehabilitation: Latarjet surgical procedure and post-operative rehabilitation.
  Interventions: Procedure: Latarjet; Other: Post-Operative Rehabilitation

INTERVENTIONS:
Procedure: Arthroscopic Bankart repair procedure — Bankart repair with remplissage consists of arthroscopic anterior inferior capsulolabral repair with arthroscopic infraspinatus tenodesis to the posterior humeral head.
  Groups: Arthroscopic Bankart repair with remplissage of Hill-Sachs lesion/rehabilitation
Procedure: Open Bankart — Open Bankart repair consists of anterior capsulorrhaphy with labral repair.
  Groups: Open Bankart/rehabilitation
Procedure: Latarjet — Latarjet consists of open transfer of the coracoid to the anterior glenoid bone deficiency.
  Groups: Latarjet/rehabilitation
Other: Post-Operative Rehabilitation — Post-operative rehabilitation will be conducted following surgical procedure-specific rehabilitation guidelines and will be progressed based on individual needs.

SUMMARY:
This clinical trial will determine the outcome trajectories of common surgeries (arthroscopic Bankart repair with remplissage of a Hill-Sachs lesion, open Bankart, Latarjet) with post-operative rehabilitation and identification of prognostic factors among patients with acute or recurrent anterior shoulder instability with subcritical bone loss. The results of the study assist in optimizing time to return to military duty, work and sports, and patient-reported physical function for military personnel and civilians with traumatic anterior shoulder instability and 10-20% glenoid bone loss. This study will provide a critical clinical advancement of a previously unaddressed and common clinical scenario.

DETAILED DESCRIPTION:
The objective of this study is to determine the outcome trajectories of common surgeries (arthroscopic Bankart repair with remplissage of a Hill-Sachs lesion, open Bankart, Latarjet) with post-operative rehabilitation and identification of prognostic factors among military personnel and civilians with acute or recurrent anterior shoulder instability with subcritical bone loss.

Aim 1: The investigators will determine the acute and long term patient relevant outcomes (Western Ontario Shoulder Instability score [WOSI], time to RTD/A at pre-injury levels, and recurrent instability/re-injury) at 6 months, 1, and 2 years of arthroscopic Bankart repair with remplissage of a Hill-Sachs lesion, open Bankart, and Latarjet.

Aim 2: The investigators will determine if participation in rehabilitation that optimizes range of motion, strength, and functional performance predicts successful RTD/A, WOSI score, and recurrent instability at 6 months, 1, and 2 years.

Subject Population: Male and female military personnel and civilians between the ages of 17 and 50 with a traumatic anterior shoulder dislocation with associated 10-20% glenoid bone loss, having undergone either an 1) arthroscopic Bankart repair with remplissage of a Hill-Sachs lesion, 2) open Bankart, or a 3) Latarjet, and plans to return to physically demanding work or sports.

Study / Experimental Design: Prospective Observational Cohort Study (Aims 1 & 2).

Methodology: Participants will undergo a standard of care computed tomography (CT) or 3D-MRI scan to quantify glenoid bone loss and shoulders with between 10-20% bone loss will be offered enrollment. We will allow shared decision-making between the patient-participant and the surgeon to occur in order to select the surgical stabilization procedure (arthroscopic Bankart repair with remplissage of a Hill-Sachs lesion, open Bankart, or Latarjet). Only those patients having one of the three surgeries will be eligible for this study. Therefore, male and female military personnel and civilians between the ages of 17 and 50 with a traumatic anterior shoulder dislocation with associated 10-20% glenoid bone loss, plans to return to physically demanding work or sports, and having undergone one of the three surgeries listed above without multi-directional instability, concomitant shoulder pathologies (e.g. rotator cuff tears, motor nerve lesion, fractures, osteoarthritis > Samilson Pietro grade 2), neuromuscular conditions including seizures, a history of shoulder surgery related to any intraarticular soft tissue, and vascular injury will be eligible to participate. We will collect information from the surgeon into what individual factors influenced the decision on surgical selection for each patient-participant.

To address the associated aims, 450 individuals will recruited and enrolled to participate in this study. Participants will be followed for 24 months, with primary outcomes consisting of patient-reported physical function and time to return to pre-injury military duty, work and sports. Secondary outcomes will include shoulder-specific and generic patient-reported measures of physical function and health related quality of life and recurrent instability.

ELIGIBILITY:
Inclusion Criteria:

* Civilians and military personnel ages 17 to 50
* Traumatic anterior shoulder dislocation
* Associated subcritical bone loss between 10-20% less the glenoid width quantified by standard of care CT scan, MRI, or 3D-MRI scan
* Had shoulder instability surgery using either 1) arthroscopic Bankart repair with remplissage of Hill-Sachs lesion; 2) open Bankart; or 3) Latarjet

Exclusion Criteria:

* Chronic, non-traumatic multi-directional instability based on clinical exam
* Concurrent shoulder injury in the involved shoulder (e.g., rotator cuff tears, motor nerve pathologies, osteoarthritis of a Samilson-Prieto grade >2)
* Have a history of shoulder surgery in the involved shoulder (prior instability surgery that included any of the following and the planned procedure would be a repeat of the index procedure: 1) arthroscopic Bankart repair with a remplissage of Hill-Sachs lesion, 2) open Bankart, or 3) Latarjet [previous isolated arthroscopic Bankart repair only would not be an exclusion criterion], rotator cuff repair, intra-articular soft tissue surgery); rotator cuff repair, intra-articular soft tissue surgery)
* Prior rotator cuff procedure on involved shoulder (including intra-articular soft tissue surgery
* Humeral sided bone lesions (Hill-Sachs lesion) that is sufficiently large enough to render the lesion "off-track" even after a bony augmentation procedure would be performed
* Neuromuscular, neurological and other movement control pathologies including seizures
* Vascular injury associated with the shoulder trauma that compromise adequate/normal healing or interferes with usual course of care
* Traumatic brain injury or any condition that would preclude the ability to comply with post-operative guidelines
* Cartilage lesion finding in the involved shoulder that would interfere with usual course of care
* Known pregnancy at time of imagining and/or surgery based upon standard of care testing procedures
* Any issue with the contralateral shoulder that would preclude participation in research procedures
* Any condition in the opinion of the investigator/clinician that would preclude or limit full participation in study activities
* Absence of a fixed address or no means of contact
* Known inability to be available at all follow-up time points
* Does not plan to return to pre-injury levels of work, sports or military duty

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female military personnel and civilians between the ages of 17 and 50 with a traumatic anterior shoulder dislocation with associated 10-20% glenoid bone loss, having undergone either an 1) arthroscopic Bankart repair with remplissage of a Hill-Sachs lesion, 2) open Bankart, or a 3) Latarjet, and plans to return to physically demanding work or sports.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability Index (WOSI) | 3 months after surgery
  The Western Ontario Shoulder Instability Index (WOSI) is a 21-item instability-specific patient-reported outcome measure of physical symptoms, sports, recreation, work, lifestyle and emotions. The best possible score is 0 and a worst possible score is 2100. The WOSI was found to be responsive and sensitive to detecting change over time, demonstrating its utility as a primary outcome to evaluate treatments and to monitor participants' progress over time.
Western Ontario Shoulder Instability Index (WOSI) | 6 months after surgery
  The Western Ontario Shoulder Instability Index (WOSI) is a 21-item instability-specific patient-reported outcome measure of physical symptoms, sports, recreation, work, lifestyle and emotions. The best possible score is 0 and a worst possible score is 2100. The WOSI was found to be responsive and sensitive to detecting change over time, demonstrating its utility as a primary outcome to evaluate treatments and to monitor participants' progress over time.
Western Ontario Shoulder Instability Index (WOSI) | 12 months after surgery
  The Western Ontario Shoulder Instability Index (WOSI) is a 21-item instability-specific patient-reported outcome measure of physical symptoms, sports, recreation, work, lifestyle and emotions. The best possible score is 0 and a worst possible score is 2100. The WOSI was found to be responsive and sensitive to detecting change over time, demonstrating its utility as a primary outcome to evaluate treatments and to monitor participants' progress over time.
Western Ontario Shoulder Instability Index (WOSI) | 24 months after surgery
  The Western Ontario Shoulder Instability Index (WOSI) is a 21-item instability-specific patient-reported outcome measure of physical symptoms, sports, recreation, work, lifestyle and emotions. The best possible score is 0 and a worst possible score is 2100. The WOSI was found to be responsive and sensitive to detecting change over time, demonstrating its utility as a primary outcome to evaluate treatments and to monitor participants' progress over time.
Time to Return to Pre-Injury Level of Activity | Monthly starting at 3 months after surgery and continuing to 24 months
  Time to return to pre-injury level military duty, work and sports.
Recurrent Instability / Re-injury | 3 months after surgery
  Recurrent instability will consist of any of the following events: dislocation, subluxation, revision stabilization procedure.
Recurrent Instability / Re-injury | 6 months after surgery
  Recurrent instability will consist of any of the following events: dislocation, subluxation, revision stabilization procedure.
Recurrent Instability / Re-injury | 12 months after surgery
  Recurrent instability will consist of any of the following events: dislocation, subluxation, revision stabilization procedure.
Recurrent Instability / Re-injury | 24 months after surgery
  Recurrent instability will consist of any of the following events: dislocation, subluxation, revision stabilization procedure.

SECONDARY OUTCOMES:
Single Assessment Numerical Evaluation (SANE) | 3 months after surgery
  The SANE is a single-item, global, patient-reported outcome measure, where the participant provides a whole number response to the question "On a scale from 0 to 100, how would you rate your injured shoulder today, with 100 being normal?" SANE scale reliability is excellent (ICC greater or equal to 0.80) and Standard Error of Measurement ranges from 4.23 to 7.82 points. Validity of the SANE displays correlations of 0.50 - 0.88 (moderate to very strong correlations) between the SANE scale and other partient-reported outcome measures.
Single Assessment Numerical Evaluation (SANE) | 6 months after surgery
  The SANE is a single-item, global, patient-reported outcome measure, where the participant provides a whole number response to the question "On a scale from 0 to 100, how would you rate your injured shoulder today, with 100 being normal?" SANE scale reliability is excellent (ICC greater or equal to 0.80) and Standard Error of Measurement ranges from 4.23 to 7.82 points. Validity of the SANE displays correlations of 0.50 - 0.88 (moderate to very strong correlations) between the SANE scale and other partient-reported outcome measures.
Single Assessment Numerical Evaluation (SANE) | 12 months after surgery
  The SANE is a single-item, global, patient-reported outcome measure, where the participant provides a whole number response to the question "On a scale from 0 to 100, how would you rate your injured shoulder today, with 100 being normal?" SANE scale reliability is excellent (ICC greater or equal to 0.80) and Standard Error of Measurement ranges from 4.23 to 7.82 points. Validity of the SANE displays correlations of 0.50 - 0.88 (moderate to very strong correlations) between the SANE scale and other partient-reported outcome measures.
Single Assessment Numerical Evaluation (SANE) | 24 months after surgery
  The SANE is a single-item, global, patient-reported outcome measure, where the participant provides a whole number response to the question "On a scale from 0 to 100, how would you rate your injured shoulder today, with 100 being normal?" SANE scale reliability is excellent (ICC greater or equal to 0.80) and Standard Error of Measurement ranges from 4.23 to 7.82 points. Validity of the SANE displays correlations of 0.50 - 0.88 (moderate to very strong correlations) between the SANE scale and other partient-reported outcome measures.
Brophy Shoulder Activity Level | 3 months after surgery
  The Brophy Shoulder Activity Level is a patient-reported measure of participant's level of sports activity. It consists of 5 items that are rated in a 5-point scale (0-4), where higher scores indicate greater activity engagement. Possible scores on the scale range from 0 - 20.
Brophy Shoulder Activity Level | 6 months after surgery
  The Brophy Shoulder Activity Level is a patient-reported measure of participant's level of sports activity. It consists of 5 items that are rated in a 5-point scale (0-4), where higher scores indicate greater activity engagement. Possible scores on the scale range from 0 - 20.
Brophy Shoulder Activity Level | 12 months after surgery
  The Brophy Shoulder Activity Level is a patient-reported measure of participant's level of sports activity. It consists of 5 items that are rated in a 5-point scale (0-4), where higher scores indicate greater activity engagement. Possible scores on the scale range from 0 - 20.
Brophy Shoulder Activity Level | 24 months after surgery
  The Brophy Shoulder Activity Level is a patient-reported measure of participant's level of sports activity. It consists of 5 items that are rated in a 5-point scale (0-4), where higher scores indicate greater activity engagement. Possible scores on the scale range from 0 - 20.
Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) - Upper Extremity (UE) | 3 months after surgery
  The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function Scale - Upper Extremity (UE) consists of an item bank of 121 items that assesses physical function regardless of the health condition present that can be administered as a computer adaptive test (CAT) or through the use of short forms. The Physical Function scale scores transformed to a T-score in which a score of 50 represents the US population average with a standard deviation of 10 indicating the population standard deviation.
Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) - Upper Extremity (UE) | 6 months after surgery
  The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function Scale - Upper Extremity (UE) consists of an item bank of 121 items that assesses physical function regardless of the health condition present that can be administered as a computer adaptive test (CAT) or through the use of short forms. The Physical Function scale scores transformed to a T-score in which a score of 50 represents the US population average with a standard deviation of 10 indicating the population standard deviation.
Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) - Upper Extremity (UE) | 12 months after surgery
  The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function Scale - Upper Extremity (UE) consists of an item bank of 121 items that assesses physical function regardless of the health condition present that can be administered as a computer adaptive test (CAT) or through the use of short forms. The Physical Function scale scores transformed to a T-score in which a score of 50 represents the US population average with a standard deviation of 10 indicating the population standard deviation.
Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) - Upper Extremity (UE) | 24 months after surgery
  The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function Scale - Upper Extremity (UE) consists of an item bank of 121 items that assesses physical function regardless of the health condition present that can be administered as a computer adaptive test (CAT) or through the use of short forms. The Physical Function scale scores transformed to a T-score in which a score of 50 represents the US population average with a standard deviation of 10 indicating the population standard deviation.
Patient-Reported Outcome Measurement Information System (PROMIS) Global-10 | 3 months after surgery
  The PROMIS-10 Global Health also measures five domains: physical function, fatigue, pain, emotional distress, and social health. Items are rated on a five-point scale. It includes physical and mental health component scores that can be transformed to t score distributions with a mean of 50 and standard deviation of 10. A higher score indicates better health.
Patient-Reported Outcome Measurement Information System (PROMIS) Global-10 | 6 months after surgery
  The PROMIS-10 Global Health also measures five domains: physical function, fatigue, pain, emotional distress, and social health. Items are rated on a five-point scale. It includes physical and mental health component scores that can be transformed to t score distributions with a mean of 50 and standard deviation of 10. A higher score indicates better health.
Patient-Reported Outcome Measurement Information System (PROMIS) Global-10 | 12 months after surgery
  The PROMIS Global-10 is a 10-item patient reported global measure of physical and emotional health. The PROMIS-10 Global Health also measures five domains: physical function, fatigue, pain, emotional distress, and social health. Items are rated on a five-point scale. It includes physical and mental health component scores that can be transformed to t score distributions with a mean of 50 and standard deviation of 10. A higher score indicates better health.
Patient-Reported Outcome Measurement Information System (PROMIS) Global-10 | 24 months after surgery
  The PROMIS Global-10 is a 10-item patient reported global measure of physical and emotional health. The PROMIS-10 Global Health also measures five domains: physical function, fatigue, pain, emotional distress, and social health. Items are rated on a five-point scale. It includes physical and mental health component scores that can be transformed to t score distributions with a mean of 50 and standard deviation of 10. A higher score indicates better health.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 3 months after surgery
  The Tampa Scale for Kinesiophobia-11 quantifies fear of re-injury due to movement and physical activity. Items are scored from 1 (strongly disagree) to 4 (strongly agree). Total TSK-11 scores range from 11 - 44, with higher scores indicating greater fear of pain, movement, and injury.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 6 months after surgery
  The Tampa Scale for Kinesiophobia-11 quantifies fear of re-injury due to movement and physical activity. Items are scored from 1 (strongly disagree) to 4 (strongly agree). Total TSK-11 scores range from 11 - 44, with higher scores indicating greater fear of pain, movement, and injury.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 12 months after surgery
  The Tampa Scale for Kinesiophobia-11 quantifies fear of re-injury due to movement and physical activity. Items are scored from 1 (strongly disagree) to 4 (strongly agree). Total TSK-11 scores range from 11 - 44, with higher scores indicating greater fear of pain, movement, and injury.
Tampa Scale for Kinesiophobia-11 (TSK-11) | 24 months after surgery
  The Tampa Scale for Kinesiophobia-11 quantifies fear of re-injury due to movement and physical activity. Items are scored from 1 (strongly disagree) to 4 (strongly agree). Total TSK-11 scores range from 11 - 44, with higher scores indicating greater fear of pain, movement, and injury.
Brief Resilience Scale | 3 months after surgery
  The Brief Resilience Scale is a 6-item questionnaire that measures an individual's ability to recover from an ongoing health related stress. It uses a 5-point Likert scale that ranges from "strongly disagree" to "strongly agree." Totally, the individual responses creates a range of possible scores from 6 - 30. The total score is then divided by the total number of questions answered for the final score. The scores range from 1 to 5, where higher scores indicate positive resilience capabilities.
Brief Resilience Scale | 6 months after surgery
  The Brief Resilience Scale is a 6-item questionnaire that measures an individual's ability to recover from an ongoing health related stress. It uses a 5-point Likert scale that ranges from "strongly disagree" to "strongly agree." Totally, the individual responses creates a range of possible scores from 6 - 30. The total score is then divided by the total number of questions answered for the final score. The scores range from 1 to 5, where higher scores indicate positive resilience capabilities.
Brief Resilience Scale | 12 months after surgery
  The Brief Resilience Scale is a 6-item questionnaire that measures an individual's ability to recover from an ongoing health related stress. It uses a 5-point Likert scale that ranges from "strongly disagree" to "strongly agree." Totally, the individual responses creates a range of possible scores from 6 - 30. The total score is then divided by the total number of questions answered for the final score. The scores range from 1 to 5, where higher scores indicate positive resilience capabilities.
Brief Resilience Scale | 24 months after surgery
  The Brief Resilience Scale is a 6-item questionnaire that measures an individual's ability to recover from an ongoing health related stress. It uses a 5-point Likert scale that ranges from "strongly disagree" to "strongly agree." Totally, the individual responses creates a range of possible scores from 6 - 30. The total score is then divided by the total number of questions answered for the final score. The scores range from 1 to 5, where higher scores indicate positive resilience capabilities.
Patient Acceptable Symptom State (PASS) | 3 months after surgery
  The Patient Acceptable Symptom State is assessed by asking the participant the question: Taking into account all the activity you have during your daily life, your level of pain and also activity limitations and participation restrictions, do you consider the current state of your shoulder satisfactory?" The PSS question is answered "Yes" or "No". A response of "Yes" indicates that the individual is satisfied with his/her current symptom state. The PASS question has show to have sufficient rest re-test reliability in patients after orthopaedic surgery, with a reported kappa coefficient of 0.78.
Patient Acceptable Symptom State (PASS) | 6 months after surgery
  The Patient Acceptable Symptom State is assessed by asking the participant the question: Taking into account all the activity you have during your daily life, your level of pain and also activity limitations and participation restrictions, do you consider the current state of your shoulder satisfactory?" The PSS question is answered "Yes" or "No". A response of "Yes" indicates that the individual is satisfied with his/her current symptom state. The PASS question has show to have sufficient rest re-test reliability in patients after orthopaedic surgery, with a reported kappa coefficient of 0.78.
Patient Acceptable Symptom State (PASS) | 12 months after surgery
  The Patient Acceptable Symptom State is assessed by asking the participant the question: Taking into account all the activity you have during your daily life, your level of pain and also activity limitations and participation restrictions, do you consider the current state of your shoulder satisfactory?" The PSS question is answered "Yes" or "No". A response of "Yes" indicates that the individual is satisfied with his/her current symptom state. The PASS question has show to have sufficient rest re-test reliability in patients after orthopaedic surgery, with a reported kappa coefficient of 0.78.
Patient Acceptable Symptom State (PASS) | 24 months after surgery
  The Patient Acceptable Symptom State is assessed by asking the participant the question: Taking into account all the activity you have during your daily life, your level of pain and also activity limitations and participation restrictions, do you consider the current state of your shoulder satisfactory?" The PSS question is answered "Yes" or "No". A response of "Yes" indicates that the individual is satisfied with his/her current symptom state. The PASS question has show to have sufficient rest re-test reliability in patients after orthopaedic surgery, with a reported kappa coefficient of 0.78.
Functional Comorbidity Index | 3 months after surgery
  The Functional Comorbidity Index (FCI) is an 18-item measure assessing the presence of medical comorbidities. The FCI is a self-administered report of medical comorbidities associated with physicla function. Using medical comorbidities is an important factor in creating risk adjustment models for orthopaedic trauma. The FCI was found to demonstrate a stronger association with the SF-36 physical function subscale (R2 = 0.29) than the Charleston (R2 = 0.18) and Kaplan-Feinstein (R2 = 0.17) indices. When individuals were classified into high and low function based ont he SF-36, the FCI correctly classified 77% of the cases.
Functional Comorbidity Index | 6 months after surgery
  The Functional Comorbidity Index (FCI) is an 18-item measure assessing the presence of medical comorbidities. The FCI is a self-administered report of medical comorbidities associated with physicla function. Using medical comorbidities is an important factor in creating risk adjustment models for orthopaedic trauma. The FCI was found to demonstrate a stronger association with the SF-36 physical function subscale (R2 = 0.29) than the Charleston (R2 = 0.18) and Kaplan-Feinstein (R2 = 0.17) indices. When individuals were classified into high and low function based ont he SF-36, the FCI correctly classified 77% of the cases.
Functional Comorbidity Index | 12 months after surgery
  The Functional Comorbidity Index (FCI) is an 18-item measure assessing the presence of medical comorbidities. The FCI is a self-administered report of medical comorbidities associated with physicla function. Using medical comorbidities is an important factor in creating risk adjustment models for orthopaedic trauma. The FCI was found to demonstrate a stronger association with the SF-36 physical function subscale (R2 = 0.29) than the Charleston (R2 = 0.18) and Kaplan-Feinstein (R2 = 0.17) indices. When individuals were classified into high and low function based ont he SF-36, the FCI correctly classified 77% of the cases.
Functional Comorbidity Index | 24 months after surgery
  The Functional Comorbidity Index (FCI) is an 18-item measure assessing the presence of medical comorbidities. The FCI is a self-administered report of medical comorbidities associated with physicla function. Using medical comorbidities is an important factor in creating risk adjustment models for orthopaedic trauma. The FCI was found to demonstrate a stronger association with the SF-36 physical function subscale (R2 = 0.29) than the Charleston (R2 = 0.18) and Kaplan-Feinstein (R2 = 0.17) indices. When individuals were classified into high and low function based ont he SF-36, the FCI correctly classified 77% of the cases.
Passive Range of Motion of the Shoulder | 3 months after surgery
  The range of passive elevation and external rotation and internal rotation of both shoulders will be measured with a goniometer. Range of motion measurements to the nearest 1 degree will be made with a large clear plastic gonionometer marked in 1 degree increments.
Passive Range of Motion of the Shoulder | 4 months after surgery
  The range of passive elevation and external rotation and internal rotation of both shoulders will be measured with a goniometer. Range of motion measurements to the nearest 1 degree will be made with a large clear plastic gonionometer marked in 1 degree increments.
Passive Range of Motion of the Shoulder | 6 months after surgery
  The range of passive elevation and external rotation and internal rotation of both shoulders will be measured with a goniometer. Range of motion measurements to the nearest 1 degree will be made with a large clear plastic gonionometer marked in 1 degree increments.
Isometric Muscle Strength of the Shoulder | 3 months after surgery
  Isometric muscle strength of shoulder will be assessed in 5 positions (external rotation at 0 degrees, external rotation at 90 degrees, internal rotation at 0 degrees, internal rotation at 90 degrees and scapular plane abduction at 90 degrees) using a hand-held dynamometer.
Isometric Muscle Strength of the Shoulder | 4 months after surgery
  Isometric muscle strength of shoulder will be assessed in 5 positions (external rotation at 0 degrees, external rotation at 90 degrees, internal rotation at 0 degrees, internal rotation at 90 degrees and scapular plane abduction at 90 degrees) using a hand-held dynamometer.
Isometric Muscle Strength of the Shoulder | 6 months after surgery
  Isometric muscle strength of shoulder will be assessed in 5 positions (external rotation at 0 degrees, external rotation at 90 degrees, internal rotation at 0 degrees, internal rotation at 90 degrees and scapular plane abduction at 90 degrees) using a hand-held dynamometer.
Performance on Functional Tests of the Upper Extremity - Closed Kinetic Chain Upper Extremity Stability test | 4 months after surgery
  Closed Kinetic Chain Upper Extremity Stability test: Participants take a full pushup position. They alternatingly touch each hand with the other, as fast as they can, for 15 seconds. Number of touches in 15 seconds.Three trials will be performed and the average value will be calculated.
Performance on Functional Tests of the Upper Extremity - Closed Kinetic Chain Upper Extremity Stability test | 6 months after surgery
  Closed Kinetic Chain Upper Extremity Stability test: Participants take a full pushup position. They alternatingly touch each hand with the other, as fast as they can, for 15 seconds. Number of touches in 15 seconds.Three trials will be performed and the average value will be calculated.
Performance on Functional Tests of the Upper Extremity - Unilateral Seated Shot-Put test | 4 months after surgery
  Unilateral Seated Shot-Put test: Distance of shot-put recorded in centimeters. The distance a 2.72 kg medicine ball is pushed, from block against participant's back to the site of ball contact on the floor. The participant will complete three trials for each arm, with the average of 3 trials being used for analysis.
Performance on Functional Tests of the Upper Extremity - Unilateral Seated Shot-Put test | 6 months after surgery
  Unilateral Seated Shot-Put test: Distance of shot-put recorded in centimeters. The distance a 2.72 kg medicine ball is pushed, from block against participant's back to the site of ball contact on the floor. The participant will complete three trials for each arm, with the average of 3 trials being used for analysis.
Performance on Functional Tests of the Upper Extremity - Push-ups | 4 months after surgery
  Push-ups: Number of push-ups that can be completed in 60 seconds is counted. The test is performed twice and the higher number of repetitions achieved is recorded.
Performance on Functional Tests of the Upper Extremity - Push-ups | 6 months after surgery
  Push-ups: Number of push-ups that can be completed in 60 seconds is counted. The test is performed twice and the higher number of repetitions achieved is recorded.
Performance on Functional Tests of the Upper Extremity - Weighted Overhead Ball Throw | 4 months after surgery
  Weighted Overhead Ball Throw: Participant will throw a 9.07 kg medicine ball overhead, with both hands. Distance of throw recorded in centimeters. Three trials will be performed.
Performance on Functional Tests of the Upper Extremity - Weighted Overhead Ball Throw | 6 months after surgery
  Weighted Overhead Ball Throw: Participant will throw a 9.07 kg medicine ball overhead, with both hands. Distance of throw recorded in centimeters. Three trials will be performed.
Performance on Functional Tests of the Upper Extremity - Upper Quarter Y-Balance test | 4 months after surgery
  Upper Quarter Y-Balance test: Maximum reach in 3 directions (medial, inferolateral, and superolateral), recorded in centimeters. Subjects stand in a three-point plank position with the tested shoulder perpendicular to the hand and the feet shoulder-width apart. Three test trials will be performed on each side with 30 seconds of rest in between each trial. A normalized composite score is the mean of the average distance in all three reach directions.
Performance on Functional Tests of the Upper Extremity - Upper Quarter Y-Balance test | 6 months after surgery
  Upper Quarter Y-Balance test: Maximum reach in 3 directions (medial, inferolateral, and superolateral), recorded in centimeters. Subjects stand in a three-point plank position with the tested shoulder perpendicular to the hand and the feet shoulder-width apart. Three test trials will be performed on each side with 30 seconds of rest in between each trial. A normalized composite score is the mean of the average distance in all three reach directions.
Clinical Measures after Surgical Stabilization - Pain | 2 weeks after surgery
  Pain: Pain intensity will be recorded utilizing an 11-point numeric pain scale (NPRS) that ranges from 0 (no pain) to 10 (worst imaginable pain). Th current, least, and worst pain intensity in the past 24 hours will be recorded and summed to create a pain score that ranges from 0 to 30.
Clinical Measures after Surgical Stabilization - Pain | 6 weeks +/- 2 weeks after surgery
  Pain: Pain intensity will be recorded utilizing an 11-point numeric pain scale (NPRS) that ranges from 0 (no pain) to 10 (worst imaginable pain). Th current, least, and worst pain intensity in the past 24 hours will be recorded and summed to create a pain score that ranges from 0 to 30.
Clinical Measures after Surgical Stabilization - Pain | 3 months after surgery
  Pain: Pain intensity will be recorded utilizing an 11-point numeric pain scale (NPRS) that ranges from 0 (no pain) to 10 (worst imaginable pain). Th current, least, and worst pain intensity in the past 24 hours will be recorded and summed to create a pain score that ranges from 0 to 30.
Clinical Measures after Surgical Stabilization - Pain | 5 months +/- month after surgery
  Pain: Pain intensity will be recorded utilizing an 11-point numeric pain scale (NPRS) that ranges from 0 (no pain) to 10 (worst imaginable pain). Th current, least, and worst pain intensity in the past 24 hours will be recorded and summed to create a pain score that ranges from 0 to 30.
Clinical Measures after Surgical Stabilization - Pain | 12 months after surgery
  Pain: Pain intensity will be recorded utilizing an 11-point numeric pain scale (NPRS) that ranges from 0 (no pain) to 10 (worst imaginable pain). Th current, least, and worst pain intensity in the past 24 hours will be recorded and summed to create a pain score that ranges from 0 to 30.
Clinical Measures after Surgical Stabilization - Pain Medication Usage | 2 weeks after surgery
  Pain Medication Usage: At follow-up visit, current narcotic pain medication usage is recorded. Usage (Yes/No): If "Yes," name of medication, dose, frequency of use, and indication is noted.
Clinical Measures after Surgical Stabilization - Pain Medication Usage | 6 weeks +/- 2 weeks after surgery
  Pain Medication Usage: At follow-up visit, current narcotic pain medication usage is recorded. Usage (Yes/No): If "Yes," name of medication, dose, frequency of use, and indication is noted.
Clinical Measures after Surgical Stabilization - Pain Medication Usage | 3 months after surgery
  Pain Medication Usage: At follow-up visit, current narcotic pain medication usage is recorded. Usage (Yes/No): If "Yes," name of medication, dose, frequency of use, and indication is noted.
Clinical Measures after Surgical Stabilization - Pain Medication Usage | 5 months +/- month after surgery
  Pain Medication Usage: At follow-up visit, current narcotic pain medication usage is recorded. Usage (Yes/No): If "Yes," name of medication, dose, frequency of use, and indication is noted.
Clinical Measures after Surgical Stabilization - Pain Medication Usage | 12 months after surgery
  Pain Medication Usage: At follow-up visit, current narcotic pain medication usage is recorded. Usage (Yes/No): If "Yes," name of medication, dose, frequency of use, and indication is noted.
Clinical Measures after Surgical Stabilization - Use of Post-op Brace | 2 weeks after surgery
  Use of Post-op Brace: Usage (Yes/No): If "No," date brace was discontinued will be recorded.
Clinical Measures after Surgical Stabilization - Use of Post-op Brace | 6 weeks +/- 2 weeks after surgery
  Use of Post-op Brace: Usage (Yes/No): If "No," date brace was discontinued will be recorded.
Clinical Measures after Surgical Stabilization - Use of Post-op Brace | 3 months after surgery
  Use of Post-op Brace: Usage (Yes/No): If "No," date brace was discontinued will be recorded.
Clinical Measures after Surgical Stabilization - Use of Post-op Brace | 5 months +/- month after surgery
  Use of Post-op Brace: Usage (Yes/No): If "No," date brace was discontinued will be recorded.
Clinical Measures after Surgical Stabilization - Use of Post-op Brace | 12 months after surgery
  Use of Post-op Brace: Usage (Yes/No): If "No," date brace was discontinued will be recorded.
Clinical Measures after Surgical Stabilization - Wound Status | 2 weeks after surgery
  Wound Status: At follow-up visit, wound status recorded as healed, healing, draining, open, erythema or presence of a superficial wound infection.
Clinical Measures after Surgical Stabilization - Wound Status | 6 weeks +/- 2 weeks after surgery
  Wound Status: At follow-up visit, wound status recorded as healed, healing, draining, open, erythema or presence of a superficial wound infection.
Clinical Measures after Surgical Stabilization - Wound Status | 3 months after surgery
  Wound Status: At follow-up visit, wound status recorded as healed, healing, draining, open, erythema or presence of a superficial wound infection.
Clinical Measures after Surgical Stabilization - Wound Status | 5 months +/- month after surgery
  Wound Status: At follow-up visit, wound status recorded as healed, healing, draining, open, erythema or presence of a superficial wound infection.
Clinical Measures after Surgical Stabilization - Wound Status | 12 months after surgery
  Wound Status: At follow-up visit, wound status recorded as healed, healing, draining, open, erythema or presence of a superficial wound infection.
Clinical Measures after Surgical Stabilization - Neurovascular status | 2 weeks after surgery
  Neurovascular status: Assessment of neurovascular status will include assessment of pulses, sensation to pain, and distal motor function. Brachial pulses will be recorded as symmetrical, diminished, or absent. Sensation to pain will be recorded as normal, diminished or absent. Distal motor function of the wrist will be recorded as strong/symmetrical to the contralateral arm, diminished, or absent.
Clinical Measures after Surgical Stabilization - Neurovascular status | 6 weeks +/- 2 weeks after surgery
  Neurovascular status: Assessment of neurovascular status will include assessment of pulses, sensation to pain, and distal motor function. Brachial pulses will be recorded as symmetrical, diminished, or absent. Sensation to pain will be recorded as normal, diminished or absent. Distal motor function of the wrist will be recorded as strong/symmetrical to the contralateral arm, diminished, or absent.
Clinical Measures after Surgical Stabilization - Neurovascular status | 3 months after surgery
  Neurovascular status: Assessment of neurovascular status will include assessment of pulses, sensation to pain, and distal motor function. Brachial pulses will be recorded as symmetrical, diminished, or absent. Sensation to pain will be recorded as normal, diminished or absent. Distal motor function of the wrist will be recorded as strong/symmetrical to the contralateral arm, diminished, or absent.
Clinical Measures after Surgical Stabilization - Neurovascular status | 5 months +/- month after surgery
  Neurovascular status: Assessment of neurovascular status will include assessment of pulses, sensation to pain, and distal motor function. Brachial pulses will be recorded as symmetrical, diminished, or absent. Sensation to pain will be recorded as normal, diminished or absent. Distal motor function of the wrist will be recorded as strong/symmetrical to the contralateral arm, diminished, or absent.
Clinical Measures after Surgical Stabilization - Neurovascular status | 12 months after surgery
  Neurovascular status: Assessment of neurovascular status will include assessment of pulses, sensation to pain, and distal motor function. Brachial pulses will be recorded as symmetrical, diminished, or absent. Sensation to pain will be recorded as normal, diminished or absent. Distal motor function of the wrist will be recorded as strong/symmetrical to the contralateral arm, diminished, or absent.
Clinical Measures after Surgical Stabilization - Additional Diagnostic Tests | 2 weeks after surgery
  Additional Diagnostic Tests: At follow-up visit, any additional diagnostic tests will be recorded. (Yes/No): If "Yes," the test, date and indication will be recorded.
Clinical Measures after Surgical Stabilization - Additional Diagnostic Tests | 3 months after surgery
  Additional Diagnostic Tests: At follow-up visit, any additional diagnostic tests will be recorded. (Yes/No): If "Yes," the test, date and indication will be recorded.
Clinical Measures after Surgical Stabilization - Additional Diagnostic Tests | 5 months +/- month after surgery
  Additional Diagnostic Tests: At follow-up visit, any additional diagnostic tests will be recorded. (Yes/No): If "Yes," the test, date and indication will be recorded.
Clinical Measures after Surgical Stabilization - Additional Diagnostic Tests | 12 months after surgery
  Additional Diagnostic Tests: At follow-up visit, any additional diagnostic tests will be recorded. (Yes/No): If "Yes," the test, date and indication will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Adam Popchak, PhD, PT, Principal Investigator — University of Pittsburgh; Jonathan Dickens, MD, Principal Investigator — Duke University; James J Irrgang, PhD, PT, Study Chair — University of Pittsburgh
Locations (15):
- United States (15):
  - Mayo Clinic, Tempe, Arizona
  - Naval Medical Center, San Diego, California
  - Steadman Clinic, Vail, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - US Naval Health Clinic (Academy), Annapolis, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital - Brown University Health, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
A public-use version of the dataset will be constructed by the Data Coordinating Center (DCC) with contents to be determined jointly by the study PIs and the DCC Director. Copies of the public-use version of the dataset will be housed at the DCC on a secure server along with suitable documentation of this dataset. The public-use version of the dataset will be exported in one or more files in simple, widely-accessible formats, e.g., .xls, .csv, and/or Statistical Analysis Software (SAS) datasets. Documentation will be in .pdf files.
Supporting Information: Study Protocol
Time Frame: The public-use version of the dataset will be made available 2 years after the study's main paper is published.
Access Criteria: Outside investigators wishing to conduct analyses using the data will submit a request with objectives, methods, and analysis plan to the PI and the Director of the DCC. Once the request is approved, the public-use version of the dataset, with documentation, will be sent by secure email using e-mail, ftp, or other mutually agreeable transmission method.